CLINICAL TRIAL: NCT06736184
Title: A Prospective Multicenter Randomized Controlled Trial on the Cardioprotective Effects of Improving Potassium Variability in Maintenance Hemodialysis Patients
Brief Title: The Cardioprotective Effects of Improving Potassium Variability in Maintenance Hemodialysis Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zunsong Wang, Chief of Nephrology Department, Qianfoshan Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: CEIPV-MHD
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Disease on Hemodialysis; Hypokalemia; Hyperkalemia; Myocardial Injury
Keywords: maintenance hemodialysis; Potassium Variability; Myocardial injury
MeSH Terms: conditions — Hypokalemia; Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potassium Variability and Myocardial Injury (Experimental)
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC)
- Control (No Intervention)

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) — 5g/meal*3meals/day
  Arms: Potassium Variability and Myocardial Injury

SUMMARY:
The management of serum potassium in maintenance hemodialysis（MHD ）patients is one of the hot topics at present. In order to control hyperkalemia in dialysis patients, the use of hypokalemic dialysate is the most important measure to reduce potassium. This measure effectively reduces serum potassium, but increases the risk of hypokalemia after dialysis, which increases the risk of all-cause death in patients. Hyperkalemia and hypokalemia during and at the end of dialysis are important factors for arrhythmia and death in MHD patients. Due to the intermittent nature of hemodialysis treatment, MHD patients often experience frequent fluctuations in serum potassium, which is a potential risk factor for poor prognosis of MHD patients. Serum potassium variability can better reflect the potassium homeostasis in MHD patients. In addition to hyperkalemia and hypokalemia, serum potassium variability is a potential risk factor affecting the prognosis of MHD patients. At present, there are few studies on the effect of improving serum potassium variability on cardiovascular complications, especially multi-center randomized controlled trials. In this study, sodium zirconium cyclosilicate was used to control hyperkalemia before dialysis and increase potassium concentration in dialysate, so as to reduce the risk of hypokalemia after dialysis, and to verify whether improving serum potassium variability can reduce myocardial injury in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Maintenance hemodialysis ≥3 months;
3. Serum potassium ≥5.0mmol/L and ≤8mmol/L before dialysis;
4. Have independent ability;
5. Complete clinical baseline data.

Exclusion Criteria:

1. Complicated with congenital heart disease, myocardial infarction and other heart diseases that may lead to cardiac dysfunction;
2. Combined with other serious diseases, such as immune diseases, severe liver and kidney dysfunction;
3. Unable to cooperate with the researcher due to mental reasons;
4. If the duration of dialysis is less than 4 hours, severe infection;
5. Patients with malignant tumors or major mental disorders;

6, except primary cardiomyopathy;

7. Severe constipation, intestinal obstruction, etc.

8. other investigators considered that enrollment was not recommended.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in QTcd at the end of dialysis in different observation groups | From enrollment to the end of treatment (totally 12 months)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pun PH, Middleton JP. Dialysate Potassium, Dialysate Magnesium, and Hemodialysis Risk. J Am Soc Nephrol. 2017 Dec;28(12):3441-3451. doi: 10.1681/ASN.2017060640. Epub 2017 Oct 9. PMID 28993507